CLINICAL TRIAL: NCT04418947
Title: Comparison of the Effectiveness of Communication Strategies on the Return to In-Person Visits to a Medical Center After the Emergence of COVID-19: A Randomized Trial
Brief Title: Project Resurgence Communication Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Anne Cappola, MD, Professor, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: 843220
Record Dates: First submitted 2020-05-29; First posted 2020-06-05 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Communication Research

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, factorial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No intervention (No Intervention)
- MPM control letter (Active Comparator)
  Interventions: Other: Communication type
- MPM intervention letter (Experimental)
  Interventions: Other: Communication type
- Mailed control letter (Active Comparator)
  Interventions: Other: Communication type
- Mailed intervention letter (Experimental)
  Interventions: Other: Communication type

INTERVENTIONS:
Other: Communication type — Control letter vs. intervention letter
  Arms: MPM control letter; MPM intervention letter; Mailed control letter; Mailed intervention letter

SUMMARY:
Randomized, double-blind, of standard of care vs additional communication and factorial design of intervention letter vs. control letter and EHR vs mail delivery mechanism in patients who canceled visits and did not reschedule over a 90 day period starting March 9, 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cancellation or failure to show for a procedure or visit from March 9, 2020 through June 7, 2020 (90 days) and who have not rescheduled as of the date of randomization

Exclusion Criteria:

* Death

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11120 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cappola AR, Schriver ER, Mowery DL, Wollack C, Ives CT, Gonzales R, Cappella JN. Effect of Targeted Messaging on Return to In-Person Visits During the COVID-19 Pandemic: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jun 1;4(6):e2115211. doi: 10.1001/jamanetworkopen.2021.15211. PMID 34190999

RESULTS

PARTICIPANT FLOW:
Groups:
- No Intervention: No letter sent to the patient
Period: Overall Study
Arm/Group | No Intervention | MPM Control Letter | MPM Intervention Letter | Mailed Control Letter | Mailed Intervention Letter
Started | 1108 | 1351 | 1351 | 3655 | 3655
Completed | 1108 | 1351 | 1351 | 3655 | 3655
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Intervention: No letter was sent to the patient.
- Total: Total of all reporting groups
Arm/Group | No Intervention | MPM Control Letter | MPM Intervention Letter | Mailed Control Letter | Mailed Intervention Letter | Total
Number analyzed (Participants) | 1108 | 1351 | 1351 | 3655 | 3655 | 11120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 627 | 797 | 797 | 2032 | 2032 | 6285
  >=65 years | 481 | 554 | 554 | 1623 | 1623 | 4835
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (6.9) | 58.4 (16.0) | 58.4 (16.2) | 59.9 (17.0) | 60.4 (17.1) | 59.7 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 609 | 757 | 756 | 1958 | 1994 | 6074
  Male | 499 | 594 | 595 | 1697 | 1661 | 5046
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 42 | 28 | 104 | 118 | 320
  Not Hispanic or Latino | 1039 | 1284 | 1298 | 3472 | 3443 | 10536
  Unknown or Not Reported | 41 | 25 | 25 | 79 | 94 | 264
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 678 | 978 | 940 | 2145 | 2089 | 6830
  Black | 291 | 259 | 273 | 1075 | 1087 | 2985
  Asian/Pacific Islander | 40 | 46 | 54 | 111 | 145 | 396
  Native American | 1 | 1 | 1 | 5 | 4 | 12
  Other | 37 | 32 | 33 | 113 | 100 | 315
  Unknown | 61 | 35 | 50 | 206 | 230 | 582
Region of Enrollment [Number; unit: participants]
  United States | 1108 | 1351 | 1351 | 3655 | 3655 | 11120

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Visit or Procedure With Provider
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention | MPM Control Letter | MPM Intervention Letter | Mailed Control Letter | Mailed Intervention Letter
Number analyzed (Participants) | 1108 | 1351 | 1351 | 3655 | 3655
Participants | 45 | 64 | 63 | 176 | 200

2. Secondary Outcome: Percent of Participants With Scheduled Visit or Procedure With Provider
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention | MPM Control Letter | MPM Intervention Letter | Mailed Control Letter | Mailed Intervention Letter
Number analyzed (Participants) | 1108 | 1351 | 1351 | 3655 | 3655
Participants | 130 | 181 | 197 | 490 | 571

3. Secondary Outcome: Percent of Participants With Completed Telemedicine Visit With Provider
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention | MPM Control Letter | MPM Intervention Letter | Mailed Control Letter | Mailed Intervention Letter
Number analyzed (Participants) | 1108 | 1351 | 1351 | 3655 | 3655
Participants | 4 | 19 | 17 | 44 | 52

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | No Intervention | MPM Control Letter | MPM Intervention Letter | Mailed Control Letter | Mailed Intervention Letter
All-Cause Mortality (participants affected / at risk) | 0/1108 | 0/1351 | 0/1351 | 0/3655 | 0/3655
Serious Adverse Events (participants affected / at risk) | 0/1108 | 0/1351 | 0/1351 | 0/3655 | 0/3655
Other Adverse Events (participants affected / at risk) | 0/1108 | 0/1351 | 0/1351 | 0/3655 | 0/3655

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT04418947/Prot_SAP_000.pdf